CLINICAL TRIAL: NCT03581981
Title: Improving Function Through Primary Care Treatment of PTSD
Brief Title: Improving Function Through Primary Care Treatment of Posttraumatic Stress Disorder (PTSD)
Acronym: PE-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency); VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2625-R
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Primary Health Care; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will not be aware of patient condition and patients will be instructed and reminded not to disclose information that may lead to unblinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged Exposure for Primary Care (PE-PC) (Experimental): Brief version of PE provided in 30 minute sessions in PC
  Interventions: Behavioral: Prolonged Exposure for Primary Care (PE-PC)
- Treatment as Usual (TAU) (Active Comparator): Veterans assigned to Primary Care (PC) Mental Health Integration (PCMHI)- Treatment as Usual (TAU) will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty Mental Health (MH)), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Prolonged Exposure for Primary Care (PE-PC) — Brief version of Prolonged Exposure (PE) provided in 30 minute sessions in primary care (PC)
  Other Names: PE-PC
  Arms: Prolonged Exposure for Primary Care (PE-PC)
Behavioral: Treatment as Usual — Veterans assigned to Primary Care (PC) Mental Health Integration (PCMHI)-Treatment as Usual (TAU) will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty MH), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
The proposed project will examine a promising brief therapy for posttraumatic stress Disorder (PTSD) for use in Veterans Health Administration (VHA) Primary Care and its impact on functional outcomes. This intervention will provide an alternative point of access to effective PTSD treatment and improved function that does not require referral to specialty mental health and accomplishes improved function in a short-term, brief protocol. Many Veterans prefer to receive mental health care, including PTSD service in primary care. The current protocol would allow them to access effective therapy options in addition to the medication management that is currently the standard of care for PTSD in primary care. In addition, this brief protocol may reduce the number of specialty mental health referrals as many Veterans may not require additional PTSD specific treatment after completion. Thus, if effective, this protocol will greatly increase Veteran treatment choice and improve functional outcomes and access while also increasing efficiency of allocation of specialty PTSD services.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a debilitating and costly mental health issue (Greenberg, Sisitsky et al. 1999, Hoge, Terhakopian et al. 2007). PTSD has an estimated two-year cost of $4.0 to $6.2 billion US dollars for mental health issues from the current conflicts in Iraq and Afghanistan and further estimated that providing evidence-based treatments for PTSD and depression could save an estimated $86.2 million (Tanielian, et al. 2008). Even modest reductions in PTSD severity have been related to increased probability of positive function outcomes (Smith, et al. 2005). Prolonged Exposure (PE) therapy (Foa, et al. 2000, Foa, et al. 2005, Schnurr, et al. 2007) is an effective, first-line treatment for PTSD (IOM 2007, VHA/Department of Defense (DOD) 2010). While highly effective, PE is provided in specialty mental health settings typically in 8 to 15, weekly 90 minute individual sessions. Veterans with PTSD are often reluctant to seek care in specialty mental health, and, as a result, many are treated solely in primary care and do not have access to this effective intervention (Possemato, et al. 2011). While the DOD and Veterans Administration (VA) have actively integrated behavioral health providers into their primary care clinics (Maguen, et al. 2010, Seal, et al. 2011), current behavioral interventions for PTSD in primary care are often inconsistent with clinical practice guidelines and/or not effective (Possemato, et al. 2011). Since functional outcomes are critical, the investigators intend to extend beyond assessing the impact of PE-PC on clinical outcomes to function. Thus, there is a clear and urgent need to further develop, validate, and disseminate evidence-based psychotherapeutic treatments for PTSD in integrated VHA Primary Care Mental Health Integration (PC-MHI) with a focus on functional outcomes. To fill this need and gap in care the study investigators developed a Brief Prolonged Exposure for Primary Care (PE-PC) treatment protocol with 4, 30-minute sessions for use in a stepped care model. A pilot study in military treatment facilities found PE-PC resulted in reductions in PTSD that were maintained at 6- and 12-month follow-up (Cigrang, et al, 2015). Preliminary results from a randomized controlled trial (RCT; PI: Cigrang; Co-Investigator: Rauch) of PE-PC compared to minimal attention control (MAC, including continuation of any PC initiated treatment) found a significantly larger reduction in PTSD severity (measured by PCL) in PE-PC than MAC (between group d = .78, p = .01). The strength of these initial findings is limited by lack of functional outcomes and examination of impact in VHA. While Service Members and Veterans have many similarities, potential differences in motivation for treatment and other factors may influence the efficacy of the protocol especially when examining changes in function. The proposed study will randomize 120 Veterans at Ralph H. Johnson Veterans Administration Medical Center (VAMC) presenting in primary care with PTSD who meet minimal inclusion/exclusion criteria to 6 weeks of PE-PC or PC-MHI-treatment as usual (TAU). Recruitment will occur over 36 months. All Veterans will complete a baseline assessment prior to randomization and post-treatment follow-up assessments at Weeks 6, 12, and 24 post-randomization. Primary outcome will be function assessed as self-reported role function in several domains. In addition, the investigators will examine symptoms severity and effectiveness, acceptability, and utilization associated with PE-PC or PCMHI-TAU in the 6 months prior to randomization and 6 months following treatment completion. PE-PC may allow access to effective treatment and efficient allocation of PTSD specialty treatment resources in the VHA. This topic is of key relevance to Veteran mental health care and can provide a new access point for high quality PTSD care to improve function allowing many more Veterans to experience improvement.

ELIGIBILITY:
Inclusion Criteria:

* Any era Veterans seeking care in VA PC for PTSD symptoms [PTSD Checklist for Diagnostic and Statistical Manual 5 (PCL-5) of at least 28)] and PTSD confirmed based on Clinician Administered PTSD Scale for Diagnostic and Statistical Manual 5 (CAPS-5)
* English speaking
* Report significant impairment in function related to PTSD symptoms as noted on intake World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
* Report that they want treatment for PTSD
* If individuals are taking psychotropic medication, 2-weeks on stable dose will be required prior to enrollment

Exclusion Criteria:

* Other primary clinical issue that would interfere with PTSD treatment
* Level of suicidal risk as determined by the Columbia Suicide Severity Rating Scale (C-SSRS) that requires:

  * PTSD + interested and consent to study
* Primary Care Provider (PCP) Screen:

  * Primary Care- Posttraumatic Stress Disorder Screen (PC-PTSD) + Intake
* PCMHI Provider:

  * [PCL 28] + brief interview

    * No PTSD OR
    * Not interested in treatment OR
    * Not interested in study
* Severe cognitive impairment that, in the judgment of the investigator, makes it unlikely that the patient can adhere to the study regimen
* Psychosis or unmanaged bipolar disorder
* Moderate to severe substance use disorder in the past 8 weeks
* Patients who are currently receiving talk therapy for trauma-related symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila A Rauch, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauch SAM, Kim HM, Acierno R, Ragin C, Wangelin B, Blitch K, Muzzy W, Hart S, Zivin K, Cigrang J. Improving function through primary care treatment of PTSD: The IMPACT study protocol. Contemp Clin Trials. 2022 Sep;120:106881. doi: 10.1016/j.cct.2022.106881. Epub 2022 Aug 12. PMID 35964868
- [Background] McLean CP, Back SE, Capone C, Morland L, Norman SB, Rauch SAM, Schnurr PP, Teng E, Acierno R. The Impact of COVID-19 on Psychotherapy Participation Among Individuals With Posttraumatic Stress Disorder Enrolled in Treatment Research. J Trauma Stress. 2022 Feb;35(1):308-313. doi: 10.1002/jts.22718. Epub 2021 Jul 22. PMID 34291832
- [Derived] Rauch SAM, Kim HM, Acierno R, Ragin C, Wangelin B, Blitch K, Muzzy W, Hart S, Zivin K. Improving function through primary care treatment of posttraumatic stress disorder study outcomes: A randomized controlled trial of prolonged exposure for primary care in veterans. Fam Syst Health. 2023 Dec;41(4):502-513. doi: 10.1037/fsh0000823. Epub 2023 Aug 31. PMID 37650808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited in VA Primary Care from April 2019 to September 2021
Pre-assignment Details: Excluded (n = 129)
  * Not meeting inclusion criteria or did not consent to study (n = 84)
  * Declined to participate (n = 45)
Groups:
- Prolonged Exposure for Primary Care (PE-PC): Brief version of Prolonged Exposure (PE) provided in 30 minute sessions in Primary Care (PC)
  Prolonged Exposure for Primary Care (PE-PC): Brief version of PE provided in 30 minute sessions in PC
- Treatment as Usual (TAU): Veterans assigned to Primary Care (PC) Mental Health Integration (PCMHI)- Treatment as Usual (TAU) will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty MH), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
  Treatment as Usual: Veterans assigned to PCMHI-TAU will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty MH), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
Period: Overall Study
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Started | 59 | 61
Completed | 46 | 42
Not Completed | 13 | 19
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Population: randomized participants
Groups:
- Prolonged Exposure for Primary Care (PE-PC): Brief version of PE provided in 30 minute sessions in PC
  Prolonged Exposure for Primary Care (PE-PC): Brief version of PE provided in 30 minute sessions in PC
- Treatment as Usual (TAU): Veterans assigned to PCMHI-TAU will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty MH), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
  Treatment as Usual: Veterans assigned to PCMHI-TAU will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty Mental Health (MH)), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (11.6) | 42.7 (14.0) | 43.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 22
  Male | 52 | 46 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 26 | 52
  Black | 31 | 30 | 61
  Other | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 61 | 120
World Health Organization Disability Assessment Scale 2.0 (WHODAS 2.0) [Mean (Standard Deviation); unit: units on a scale] — WHODAS is a 36-item disability interviewer administered assessment covering six domains of function: cognition, mobility, self-care, getting along, life activities, and participation. Each item is scored as none, mild, moderate, severe, or extreme/cannot do. Simple scoring where items are summed across the scale was used. Total scores can range from range from 0 (no disability) to 144 (full disability) with higher scores indicate greater functional impairment.
  units on a scale | 48.8 (18.1) | 46.7 (16.1) | 47.7 (17.1)
Clinician Administered PTSD Scale for Diagnostic and Statistical Manual 5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — CAPS-5 is a 30 -item interviewer administered assessment of PTSD severity over the past month. Each item is scored as absent, mild/subthreshold, moderate/threshold, severe/markedly elevated, or extreme/incapacitating and summed for the total score. The scores ranges from 0 to 80 higher as more severe PTSD. Clinical cut scores for interpretation of this measure have not yet been established..
  units on a scale | 34.0 (8.8) | 34.1 (9.3) | 34.0 (9.0)
Patient Health Questionnaire 9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — PHQ-9 is a 9 item self-report measure of depressive symptoms over the past two weeks. Each item is scored as not at all, several days, more than half days, or nearly every day and summed for the total score. Scores range from 0 (no depression) to 27 (most severe depression). Higher scores would be more severe depression and 10 and higher is considered depressed. Total scores are interpreted as: Minimal 1-4; Mild 5-9; moderate 10-14; Moderately sever 15-19; Severe 20+
  units on a scale | 14.1 (5.1) | 15.0 (5.5) | 14.6 (5.3)
PTSD Checklist for Diagnostic and Statistical Manual 5(PCL-5) [Mean (Standard Deviation); unit: units on a scale] — PCL-5 is a 20 item self-report assessment of the PTSD symptoms over the past month. Each item is scored as not at all, a little bit, moderately, quite a bit, or extremely and summed for the total score. The scores ranges from 0 to 80 higher as more severe PTSD. PCL-5 cutoff score between 31-33 is indicative of probable PTSD.
  units on a scale | 49.4 (11.6) | 50.9 (13.0) | 50.1 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Disability Assessment Scale 2.0 Change
Description: Change in total score between Week 6 and Week 0 time points can range from 144 (total disability after full function) to 0 (no change) to -144 (total recovery of all function after total disability). Lower change scores reflect more return of function between timepoints. Cut points for this measure have not yet been established.
Time Frame: Week 6 to Week 0
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment as Usual (TAU): Veterans assigned to PCMHI-TAU will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty MH), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
  Treatment as Usual: Veterans assigned to PCMHI-TAU will receive standard PCMHI care for PTSD in PC that does not include any PTSD-specific therapy in PCMHI but may include referral for specialty care (including specialty MH), medication management or general supportive contact while awaiting referral. All PTSD care received during the study will be collected and monitored as TAU.
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 43 | 50
units on a scale | -7.5 (21.3) | -4.3 (14.9)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority — see statistical plan; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-10.7 to 3.6]

2. Primary Outcome: World Health Organization Disability Assessment Scale 2.0
Description: WHODAS is a 36-item disability interviewer administered assessment covering six domains of function: cognition, mobility, self-care, getting along, life activities, and participation. Each item is scored as none, mild, moderate, severe, or extreme/cannot do. Simple scoring where items are summed across the scale was used. Total scores can range from range from 0 (no disability) to 144 (full disability) with higher scores indicate greater functional impairment.
Time Frame: Week 12
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 48 | 42
units on a scale | 56.9 (28.8) | 51.5 (24.1)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Final Values) = 0.61

3. Primary Outcome: World Health Organization Disability Assessment Scale 2.0
Description: as for outcome 2
Time Frame: Week 24
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 46 | 42
units on a scale | 58.1 (29.7) | 53.9 (28.3)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Final Values) = 0.61

4. Secondary Outcome: Clinician Administered PTSD Scale for Diagnostic and Statistical Manual 5 (CAPS-5) Change
Description: Change scores range between Week 6 and Week 0 time points from 80 (Most severe PTSD after no PTSD) to 0 (no change) to -80 (No PTSD after most severe PTSD). Lower change score indicates more reduction in PTSD. Cut points for this change measure have not yet been established.
Time Frame: Week 6 to Week 0
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 43 | 50
units on a scale | -3.4 (11.1) | -3.1 (7.4)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-3.6 to 3.6]

5. Secondary Outcome: PTSD Checklist for Diagnostic and Statistical Manual 5 (PCL-5) Change
Description: as for outcome 4
Time Frame: Week 6 to Week 0
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 41 | 48
units on a scale | -6.9 (18.1) | -5.7 (7.7)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-7.3 to 3.7]

6. Secondary Outcome: Patient Health Questionnaire- 9 (PHQ-9) Change
Description: Change scores range between Week 6 and Week 0 time points from 27 (Most severe depression after no depression) to 0 (no change) to -27 (No depression after most severe depression). Lower change score indicates more reduction in depression. Cut points for this change measure have not yet been established.
Time Frame: Week 6 to week 0
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 41 | 47
units on a scale | -1.1 (5.9) | -2.0 (4.4)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.50, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.4 to 2.9]

7. Secondary Outcome: Clinician Administered PTSD Scale for Diagnostic and Statistical Manual 5 (CAPS-5)
Description: CAPS-5 is a 30 -item interviewer administered assessment of PTSD severity over the past month. Each item is scored as absent, mild/subthreshold, moderate/threshold, severe/markedly elevated, or extreme/incapacitating and summed for the total score. The scores ranges from 0 to 80 higher as more severe PTSD. Clinical cut scores for interpretation of this measure have not yet been established.
Time Frame: Week 12
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 48 | 42
units on a scale | 28.8 (14.0) | 28.4 (11.2)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 0.00

8. Secondary Outcome: Clinician Administered PTSD Scale for Diagnostic and Statistical Manual 5 (CAPS-5)
Description: as for outcome 7
Time Frame: Week 24
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 46 | 42
units on a scale | 28.1 (12.7) | 28.6 (11.8)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 0.00

9. Secondary Outcome: PTSD Checklist for Diagnostic and Statistical Manual 5 (PCL-5)
Description: PCL-5 is a 20 item self-report assessment of the PTSD symptoms over the past month. Each item is scored as not at all, a little bit, moderately, quite a bit, or extremely and summed for the total score. The scores ranges from 0 to 80 higher as more severe PTSD. PCL-5 cutoff score between 31-33 is indicative of probable PTSD.
Time Frame: Week 12
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 47 | 38
units on a scale | 41.1 (20.4) | 40.2 (15.6)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Final Values) = 1.45

10. Secondary Outcome: PTSD Checklist for Diagnostic and Statistical Manual 5 (PCL-5)
Description: as for outcome 9
Time Frame: Week 24
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 44 | 39
units on a scale | 42.1 (20.5) | 40.5 (16.6)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Final Values) = 1.45

11. Secondary Outcome: Patient Health Questionnaire- 9 (PHQ-9)
Description: PHQ-9 is a 9 item self-report measure of depressive symptoms over the past two weeks. Each item is scored as not at all, several days, more than half days, or nearly every day and summed for the total score. Scores range from 0 (no depression) to 27 (most severe depression). Higher scores would be more severe depression and 10 and higher is considered depressed. Total scores are interpreted as: Minimal 1-4; Mild 5-9; moderate 10-14; Moderately sever 15-19; Severe 20+
Time Frame: Week 12
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 47 | 38
units on a scale | 12.5 (6.8) | 12.8 (5.9)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.41, Mixed Models Analysis; Mean Difference (Final Values) = 2.87

12. Secondary Outcome: Patient Health Questionnaire- 9 (PHQ-9)
Description: as for outcome 11
Time Frame: Week 24
Population: All those with 4 or fewer missing items on the measure are included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
Number analyzed (Participants) | 44 | 39
units on a scale | 13.1 (6.6) | 12.2 (5.9)
Statistical Analysis 1: Comparison: Prolonged Exposure for Primary Care (PE-PC) vs Treatment as Usual (TAU); Test type: Superiority; p = 0.41, Mixed Models Analysis; Mean Difference (Final Values) = 2.87

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events were collected at each clinical or assessment contact.
Arm/Group | Prolonged Exposure for Primary Care (PE-PC) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/61
Other Adverse Events (participants affected / at risk) | 0/59 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure for Primary Care (PE-PC) (N=59) | Treatment as Usual (TAU) (N=61)
Attempted Suicide (Psychiatric disorders) | 1 (1) | 0 (0) — patient with history of attempting suicide attempted by pill overdose and contacted others for help. patient was hospitalized and removed from the study and provided care. Outside study providers and review indicated not related to the study.

LIMITATIONS AND CAVEATS:
Note that the 2 PCMHI clinics in the current study employ primarily cognitive behavioral therapies (e.g., exposure, behavioral activation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03581981/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03581981/ICF_001.pdf